CLINICAL TRIAL: NCT02709408
Title: Prospective Observational Study to Assess the Risk Factors, Clinical Management and Outcomes of Hospitalized Patients With Serious Infections Caused by Carbapenem-resistant Enterobacteriaceae and Acinetobacter Baumannii
Brief Title: European Prospective Cohort Study on Enterobacteriaceae Showing Resistance to Carbapenems
Acronym: EURECA
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: COMBACTE-CARE WP1A
Record Dates: First submitted 2016-03-02; First posted 2016-03-16 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Carbapenem Resistant Bacteria Infection
Keywords: Carbapenem resistance; Enterobacteriaceae; Acinetobacter baumannii; Bloodstream infections; Intrabdominal infections; Urinary tract infections; Pneumonia; Risk factors; Outcome; Hospitalised patients; Mortality; Clinical response; Length of hospital stay
MeSH Terms: conditions — Sepsis; Urinary Tract Infections; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Bacteria (carbapenem-resistant and susceptible Enterobacteriaceae, carbapenem-resistant Acinetobacter baumannii)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Carbapenem-resistant Enterobacteriaceae: Patients with complicated intrabdominal infections, pneumonia, complicated urinary tract infection and bloodstream infection due to carbapenem-resistant Enterobacteriaceae
- Carbapenem-resistant A. baumannii: Patients with bloodstream infections due to carbapenem-resistant Acinetobacter baumannii
- Susceptible Enterobacteriaceae: Patients with complicated intrabdominal infections, pneumonia, complicated urinary tract infection and bloodstream infection due to carbapenem-susceptible Enterobacteriaceae matched to carbapenem-resistant ones by centre, type of ward, infection type, acquisition and previous duration of hospitalisation.
- Admitted control patients: Patients without infection due to Enterobacteriaceae matched to carbapenem-resistant Enterobacteriaceae cases according to centre, ward and previous length of hospitalisation.

SUMMARY:
Among antibiotic-resistant organisms, the Gram-negative bacteria are now the most important challenge because of the rapid worldwide spread of mechanisms conferring resistance to multiple drugs. The most recent and worrying problem is the emergence and spread of carbapenemases. Additionally, carbapenem-resistance is known to be very frequent among Acinetobacter baumannii isolates for many years. Overall, the therapeutic options available against carbapenem-resistant Enterobacteriaceae (CRE) and A. baumannii (CRAB) are very limited. The best available treatment (BAT) against CRE is unknown, which is a challenge for therapeutic decisions and also for the design of randomized trials with new drugs. The generic objectives of EURECA are to obtain high-quality observational data to inform the design of randomized controlled trials for complicated intraabdominal infections, pneumonia, complicated urinary tract infections and bloodstream infections due to Carbapenem-resistant Enterobacteriaceae (CRE) and carbapenem-resistant Acinetobater baumannii, and to provide cohort data that could eventually be used as historical controls for future comparisons with new drugs targeting CRE. This will be achieved by a prospective, multinational cohort study of patients with targeted infections due to CRE and CRAB, and by matched case-control-control studies.

DETAILED DESCRIPTION:
HYPOTHESIS:

H1: 5 independent predictors for cure and mortality can be identified, including active empirical therapy, early targeted optimized therapy and early source management if needed.

H2: For pneumonia, cIAI (complicated intrabdominal infection) and BSI (bloodstream infection), combination therapy with two active drugs, one of them being (if available) an "active" beta-lactam (such as meropenem or imipenem if minimum inhibitory concentration [MIC] <16 mg/L, aztreonam if isolate is susceptible as in many metallo-beta-lactamase producers, or cephalosporin if isolate is susceptible as in some OXA-48 producers). For cUTI (complicated urinary tract infection), monotherapy with an "active" beta-lactam as above, colistin or an aminoglycoside (if active in vitro) is as effective as combination therapy.

H3. Clinical cure rate at test of cure (TOC) will be 50% with BAT. H4: Specific carbapenemase types do not independently influence cure rate or mortality.

H5: CRE infections caused by isolates showing a carbapenem MIC <16 mg/L are associated with higher probability of cure and lower mortality.

H6: five significant independent predictors (risk factors) for CRE infection can be found.

H7: the targeted infections due to CRE are significantly and independently associated with higher mortality, hospital stay and hospital costs than infections caused by carbapenem-susceptible Enterobacteriaceae (CSE) or than other diseases causing hospitalisation.

SPECIFIC OBJECTIVES. O1. To characterise the features, clinical management and outcomes of hospitalised patients with cIAI, pneumonia, cUTI and BSI caused by CRE and CRAB.

O1A. To provide cohorts of patients with the targeted infections caused by CRE and CRAB that would eventually be used as historical cohorts for comparison of efficacy and safety of newer drugs against these organisms.

O1B. To identify the outcome predictors of patients with cIAI, pneumonia, cUTI and BSI caused by CRE and CRAB, with identification of the best alternative therapy (BAT).

O1C. To exploratively investigate the importance of the specific carbapenemase and carbapenem-MIC in the outcome of CRE and CRAB infections.

O2. To identify the risk factors for target infections caused by CRE to inform a more efficient design of future randomized clinical trials for these infections.

O3. To assess the mortality, length of hospital stay and hospital costs associated with target infections caused by CRE.

DESIGN AND STUDIES To answer the above objectives, a prospective, multinational, multicentre, observational and analytic project including 3 studies was design.

Study 1. For the analysis of outcome predictors of CRE and CRAB infections (objective 1), a prospective cohort study of patients with the target infections due to CRE and CRAB will be performed.

Study 2. For the analysis of risk factors for target infections caused by CRE (objective 2), a nested case-control-control will be performed. The first group of controls will be formed by matched patients with CSE infections, and the second groups of controls will be formed by admitted patients non-infected patients by CRE or CSE.

Study 3. For the analysis of cost, outcome impact and length of stay associated to target infections caused by CRE (objective 3), a matched cohorts study will be performed. The cohorts will be formed by selected patients with infections due to CRE and the patients with infections due to CSE (identical to the CSE control group above). Additionally, a control group of admitted patients not infected by CRE or CSE will be studied (identical to the admitted control group above).

SETTING This study will be performed in 50 European hospitals from Spain, Italy, Greece, Turkey, Serbia, Croatia, Montenegro, Kosovo, Albania, Bulgaria and Romania.

STUDY PERIOD The recruitment period of the study is planned from February 2016 to June 2017.

ENDPOINTS (MAIN OUTCOME VARIABLES) See below

STUDY VARIABLES AND DEFINITIONS

* CRE: any isolate identified as an Enterobacteriaceae showing a minimum inhibitory concentration (MIC) ≥1 mg/L if using any dilution method and/or ≤22 mm if using a disc-diffusion method for imipenem or meropenem (10 µg disks); all others will be considered carbapenem susceptible (CSE), but meropenem and imipenem susceptible isolates showing resistance to ertapenem will be excluded.
* CRAB: Any isolate identified as Acinetobacter baumannii showing a minimum inhibitory concentration (MIC) ≥16 mg/L for imipenem or meropenem if using any dilution method and/or ≤17 mm for meropenem and/or ≤15 for imipenem if using a disc-diffusion method.
* Independent variables for Study 1: demographics, comorbidities in adults (Charlson's index), comorbidities in children (ARPEC PPS definitions), type of acquisition, systemic inflammatory response syndrome severity in adults, sepsis criteria in children, Pitt score, SOFA score, APACHE-II score, PIM2, invasive procedures, neutropenia, microbiological variables (poly or monomicrobial infection, carbapenemase producer, carbapenemases type, susceptibility profile, carbapenem MIC), clinical management (source control and support therapy), antimicrobial therapy.
* Independent variables for Study 2: demographics, length of hospital stay, epidemiological variables (travels, previous contact with persons colonised by CRE, previous hospitalization, nursing home or other long term-care facility residency, previous colonisation by CRE), comorbidities, acquisition type, SIRS severity in adults, sepsis in children, Pitt score, SOFA score, APACHE-II score, PIM2, invasive procedures, neutropenia, type of infection, microbiological variables, antibiotics received in the last 3 months.
* Independent variables for Study 3: all those included in Study 2.

DATA COLLECTION AND FOLLOW-UP Data will be collected by trained local investigators. Patients will be followed for 30 days from day 0. Data prior to study entry will be collected by reviewing medical records or interviewing the patient, his/her family or the attending healthcare staff. After that, the patients will be followed prospectively. If the patients had been discharged before assessement, outcome must be assessed by an outpatient visit or phone call according to a pre-design questionnaire.

MICROBIOLOGICAL STUDIES. All procedures will be performed locally using accepted, standard microbiological protocols. Isolates identified as CRE or CRAB according to above criteria will be locally studied for carbapenemase production using the CARBA-NP test. Susceptibility tests to key antimicrobial agents will be collected. Isolates preservation CRE and CRAB isolates will be preserved locally at least at -20ºC.

SAFETY ASSESMENT No investigation drugs will be used in this study. Adverse event will be collected during follow-up as one variable of interest for analysis purposes.

SAMPLE SIZE :

* Study 1 The sample size for the CRE and CRAB cohorts were calculated so that the cohorts may serve as 'historical' cohorts for future comparison with new drugs for CRE and CRAB. To do so, and because the estimates for the outcome variable of the new drug is unknown, we seek to estimate the clinical cure rate of BAT with 95% confidence interval and 8% precision. For an estimated cure rate of 50% based on data from previous studies, 151 patients for each of the five types of infection are needed (due to CRE: cUTI, pneumonia, cIAI, and BSI; due to CRAB: BSI). However, because around 25% of patients will not receive BAT, we will need 201 patients per type of infection except for BSI due to A. baumannii, for which we will need 221 because some blood isolates identified as Acinetobacter spp in sites not specifying the species will not be A. baumannii (total, 1025 patients). Such sample size will be enough also to investigate the best available therapy with the merged CRE cohorts.
* Study 2: The CRE case group will be formed by 248 patients with CRE infections selected from the study 1 cohort. Per each CRE case, one CSE control patient and 3 non-infected controls will be selected. Because of possible heterogeneity due to the different infection types, we have chosen to over sample by a ratio of 248/201*100%. The number of matched controls has been chosen to be four which is well known to well approximate the power of full cohort data.
* Study 3 The CRE, CSE and non-infected cohorts will be formed by the same patients as in Study 2. Therefore, the sample size rationale is as for Study 2, however with the refinement that the nested case control matching is now viewed as an exposure density sampling.

STATISTICAL ANALYSIS

* Study 1. The outcomes associated with exposure to different variables will be compared; the targeted exposures will be empirical active antimicrobial therapy, early targeted optimized therapy, and early source control. Antimicrobial regimens will be analysed as empirical (administered before the susceptibility testing is available) and targeted (thereafter) therapy. The primary endpoint "mortality from any cause until day 30" will be analysed using survival methods (Kaplan-Meier, Cox regression). The other primary endpoint "clinical response at TOC" will be analysed as a dichotomous outcome, regression analyses will use the logistic regression model. The analysis of the secondary endpoints will be analogous. Microbiological response at TOC is a polychotomous outcome and will be analysed using multinomial logistic regression. Goodness of fit will be assessed throughout. Variable selection will be based on Akaike's information criterion.
* Study 2. Exposure to potential risk factors of patients will be compared between CRE cases and CSE controls, and between CRE cases and admitted controls. A stratified and weighted Cox analysis will be performed. Multilevel hospital data (local rate of CRE, antimicrobial consumption, infection control measures) will also be considered in the analyses above.
* Study 3. The impact of CRE infection on mortality, length of stay, cost, length of hospital and ICU stay, and length of mechanical ventilation of patients will be assessed by comparison with those of CSE infection and admitted patients. All time-to-event outcomes (for costs and extra hospital/ICU days see below) will be compared using survival techniques. Because the outcome infection due to CRE is subject to the competing risks of death in hospital w/o CRE infection and discharged alive from hospital with or without CRE infection, the analyses shall be supplemented by those of the competing outcomes. Goodness of fit will be assessed throughout. Extra hospital/ICU days will be estimated using the multistate approach of Beyersmann et al. Variable selection will be based on Akaike's information criterion. Goodness of fit will be assessed throughout.

ETHICAL CONSIDERATIONS. Prior to initiation of a study site, approval will be sought from the appropriate regulatory agency and local Ethics Committees of Research or IRBs to conduct the study in accordance with regulatory requirements. This is an observational study and therefore no intervention is performed on behalf of the investigation. Management of all patients including all antibiotic regimens prescribed will be decided by the physician doctor/team in charge without any interference. The processing of the patients' personal data collected in this study shall comply with the Data Protection Act 1998 and with the European Directive on the Privacy of Data.

MONITORING The study will be monitored for quality and consistency of data.

ELIGIBILITY:
Selection criteria for CRE GROUPS and CRAB GROUP:

Inclusion criteria (all must be fulfilled):

* Isolation of CRE or CRAB from a clinical sample (e.g., a sample obtained in the work-up of a patient with suspicion of infection; therefore, screening samples are not considered).
* The patient meets the criteria for any of the following infections (see definitions below): complicated urinary tract infection, pneumonia, intraabdominal infection or bloodstream infection (if the source of infection is any of the above, the patient will be included in both groups).
* Patient or his/her representative sign the inform consent if requested by the local Institutional Review Board (IRB).

Patients in these groups will be included until the needed sample sizes are reached.

Exclusion Criteria:

* The infection is considered to be polymicrobial according to standard microbiological interpretation of culture results (except for cIAI, in which polymicrobial infections are allowed).
* The patient was participating in a clinical trial that involved active treatment for the infections.
* The patient was previously included in the same cohort of this study for the same organism. A single episode of CRE or CRAB per patient can be included. Patients who suffer a CRE infection could later be included in the CRAB cohort if developing a CRAB infection and vice versa.
* Patients with do not resuscitate orders or with a life expectancy of <30 days. Selection criteria for CSE GROUP Inclusion criteria (all must be fulfilled)
* Isolation of CSE from a clinical sample (e.g., a sample obtained in the work-up of a patient with suspicion of infection; therefore, screening samples are not considered).
* The patient meets the criteria for any of the following infections (see definitions below): complicated urinary tract infection, pneumonia, intraabdominal infection or bloodstream infection (if the source of infection is any of the above, the patient will be included in both groups).
* The infection is the same as that of the index case; in case of BSI, the source of bacteraemia must be the same as the index case classified as follows: UTI, pneumonia, intraabdominal infection or any other.
* The type of acquisition is the same as for the index CRE case (nosocomial or community).
* The previous length of hospitalization before the infection onset is minus 1 up to minus 3 days the previous length of hospitalization before the CRE infection date in the CRE correspondent (up to minus 7 days if the CRE case occurred after 14 days of previous stay).
* The patient was admitted to the same type of service as the index case (medical, surgical, ICU, neonatal Unit, paediatric ICU, general paediatric wards).
* Patient or his/her representative sign the inform consent (if requested by local IRB).

Patients in this group will be included until the needed sample size is reached.

Exclusion criteria

* The infection is considered to be polymicrobial according to standard microbiological interpretation of culture results (except for cIAI, in which polymicrobial infections are allowed).
* Patient is participating in a clinical trial that involved active treatment for the infections at assessment.
* Patients with do not resuscitate orders or with a life expectancy of <30 days. The first patient found with all inclusion criteria and no exclusion criteria will be included.

Selection criteria for ADMITTED CONTROL GROUP Inclusion criteria (all must be fulfilled)

* Patient is admitted in the same hospital ward where was admitted the index CRE.
* The previous length of hospitalization is at least one day less than the previous duration of hospitalisation of the correspondent CRE case when the CRE infection occurred.
* Patient or his/her representative sign the inform consent (if requested by local IRB).

Patients in this group will be included until the needed sample size is reached.

Exclusion criteria

* Patient was participating in a clinical trial that involved active treatment for the infections at assessment.
* Patients with do not resuscitate orders or with a life expectancy of <30 days.

Because the search for CSE controls is more difficult, the search for admitted control patients can be started once a CSE control has been included; the first 3 patients with the above inclusion criteria and no exclusion criteria will be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The base-population for the studies are:
  * Study 1: all patients with the targeted infections due to CRE or CRAB.
  * Study 2 and study 3: all admitted patients with the targeted infections due to CRE or CSE, and all admitted patients.
Sampling Method: Non-Probability Sample
Enrollment: 2515 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Death by any caused
Clinical response (failure vs cure or improvement) | 21 days
  Clinical failure: non-improvement or deterioration (clinical situation qualified as similar or worse in comparison to that at the diagnosis of bacteremia), death (death of the patient for whatever the reason) or relapse (reappearance of signs and symptoms related to the infection, after the end of treatment).
  Clinical cure: resolution of all signs and symptoms related to the infection, and antibiotic therapy is no longer necessary.
  Clinical improvement: resolution or partial improvement of signs or symptoms of the infection at the time of assessment but antibiotic therapy is still needed.
  TOC was decided at day 21 because it is usually 7 days after the expected average duration of therapy, which is around 10-14 days for the infections included.
Infection due to CRE | 1 year
  Infection due to CRE (study 2)
Length of hospital stay. | 1 year
  Duration of hospitalisation (study 3)

SECONDARY OUTCOMES:
Microbiological response (microbiological eradication, failure or uncertain). | 21 days
  Microbiological eradication: follow-up cultures from the infection site are negative for the causative pathogen; if follow-up cultures were not performed for clinical reasons but there is clinical cure, the case is classified as "microbiological eradiation, presumptive".
  Microbiological failure: follow-up cultures from the infection site are still positive for the causative pathogen.
  Uncertain: follow-up cultures were not performed but there is no clinical cure.
Mortality during hospitalisation. | 1 year
  Death from any cause only during the hospitalisation of the patient.
Infection-related mortality | 30 days
  Death occurring in direct relation to the infection or its complications, and without any other alternative reasonable explanation, in opinion of the local investigator.
Length of hospital stay after the infection (and ICU stay, mechanical ventilation if appropriate). | After end of hospitalisation
  Duration of hospitalisation (and in ICU or of mechanical ventilation if appropriate).
Duration of antibiotic treatment for the episode. | 30 days
  Days of antibiotic therapy for the infection
Recurrence | 30 days
  Reappearance of infection by the same organism.
Superinfection | 30 days
  Occurrence of any infection by a different organism.
Therapy-related adverse events. | 30 days
  Moderate to severe adverse events related to treatment of the infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rodríguez Baño, MD, PhD, Study Chair — FISEVI (Fundación Pública Andaluza para la Gestión de la Investigación en Salud de Sevilla
Locations (50):
- Spitali i Sanatoriumit Shefqet Ndroqi, Tirana, Albania
- Meditsinski Center-N.I Pirogov, Totleben, Bulgaria
- University Hospital for Infectious Diseases, Zagreb, Croatia
- Greece (10):
  - Agioi Anargyroi General Hospital of Athens, Athens
  - Attikon University Hospital, Athens
  - Evangelismos General Hospital of Athens, Athens
  - Laiko General Hospital, Athens
  - Iaso General Hospital, Cholargós
  - General Hospital of Larissa, Larissa
  - General University Hospital of Larissa, Larissa
  - General University Hospital of Patras, Pátrai
  - Hippokration General Hospita, Thessaloniki
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
- Italy (10):
  - Policlinico S. Orsola Malpighi, Bologna
  - Florence University Hospital, Florence
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Hospital Luigi Sacco, Milan
  - University of Milan-Bicocca, San Gerardo, Milan
  - University of Naples S.U.N./Monaldi Hospital, Naples
  - San Martino University Hospital, Padua
  - National Institute for Infectious Diseases Lazzaro Spallanzani, Rome
  - Policlinico Universitario A. Gemelli, Rome
  - Molinette Teaching Hospital, Torino
- University Clinical Center of Kosovo, Pristina, Kosovo
- Clinical Center of Montenegro, Podgorica, Montenegro
- Romania (7):
  - Elias Emergency University Hospital, Bucharest
  - Fundeni Clinical Hospital, Bucharest
  - Infectious and Tropical Diseases Hospital "Dr. Victor Babes", Bucharest
  - The National Institute for Infectious Diseases "Prof. Dr. Matei Bals", Bucharest
  - Cluj-Napoca Infectious diseases Clinical Hospital, Cluj-Napoca
  - Clinical Hospital of Infectious Diseases of Iasi, Iași
  - The Mures County Clinical Emergency Hospital, Târgu Mureş
- Serbia (5):
  - Clinical Center of "Dragisa Misovic", Belgrade
  - Clinical Centre of Serbia, Belgrade
  - Clinical Center Nis, Niš
  - Clinical Centre of Vojvodina, Novi Sad
  - University Clinical Center Zvezdara, Zvezdara
- Spain (8):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Gregorio Marañón, Madrid
  - Hospital Puerta del Hierro, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Carlos Haya, Málaga
- Turkey (Türkiye) (5):
  - Ankara University, Ankara
  - Hacettepe University School of Medicine, Ankara
  - Uludağ University, Bursa
  - Marmara University, Istanbul
  - Izmir Chest Diseases and Surgery Training and Research Hospital, Konak

IPD SHARING:
Plan to Share IPD: Yes
Within COMBACTE consortium

REFERENCES:
- [Background] Tzouvelekis LS, Markogiannakis A, Psichogiou M, Tassios PT, Daikos GL. Carbapenemases in Klebsiella pneumoniae and other Enterobacteriaceae: an evolving crisis of global dimensions. Clin Microbiol Rev. 2012 Oct;25(4):682-707. doi: 10.1128/CMR.05035-11. PMID 23034326
- [Background] Grundmann H, Livermore DM, Giske CG, Canton R, Rossolini GM, Campos J, Vatopoulos A, Gniadkowski M, Toth A, Pfeifer Y, Jarlier V, Carmeli Y; CNSE Working Group. Carbapenem-non-susceptible Enterobacteriaceae in Europe: conclusions from a meeting of national experts. Euro Surveill. 2010 Nov 18;15(46):19711. doi: 10.2807/ese.15.46.19711-en. PMID 21144429
- [Background] Tumbarello M, Viale P, Viscoli C, Trecarichi EM, Tumietto F, Marchese A, Spanu T, Ambretti S, Ginocchio F, Cristini F, Losito AR, Tedeschi S, Cauda R, Bassetti M. Predictors of mortality in bloodstream infections caused by Klebsiella pneumoniae carbapenemase-producing K. pneumoniae: importance of combination therapy. Clin Infect Dis. 2012 Oct;55(7):943-50. doi: 10.1093/cid/cis588. Epub 2012 Jul 2. PMID 22752516
- [Background] Qureshi ZA, Paterson DL, Potoski BA, Kilayko MC, Sandovsky G, Sordillo E, Polsky B, Adams-Haduch JM, Doi Y. Treatment outcome of bacteremia due to KPC-producing Klebsiella pneumoniae: superiority of combination antimicrobial regimens. Antimicrob Agents Chemother. 2012 Apr;56(4):2108-13. doi: 10.1128/AAC.06268-11. Epub 2012 Jan 17. PMID 22252816
- [Background] Daikos GL, Tsaousi S, Tzouvelekis LS, Anyfantis I, Psichogiou M, Argyropoulou A, Stefanou I, Sypsa V, Miriagou V, Nepka M, Georgiadou S, Markogiannakis A, Goukos D, Skoutelis A. Carbapenemase-producing Klebsiella pneumoniae bloodstream infections: lowering mortality by antibiotic combination schemes and the role of carbapenems. Antimicrob Agents Chemother. 2014;58(4):2322-8. doi: 10.1128/AAC.02166-13. Epub 2014 Feb 10. PMID 24514083
- [Background] Paul M, Carmeli Y, Durante-Mangoni E, Mouton JW, Tacconelli E, Theuretzbacher U, Mussini C, Leibovici L. Combination therapy for carbapenem-resistant Gram-negative bacteria. J Antimicrob Chemother. 2014 Sep;69(9):2305-9. doi: 10.1093/jac/dku168. Epub 2014 May 28. PMID 24872346
- [Background] Rodriguez-Bano J, Cisneros JM, Cobos-Trigueros N, Fresco G, Navarro-San Francisco C, Gudiol C, Horcajada JP, Lopez-Cerero L, Martinez JA, Molina J, Montero M, Pano-Pardo JR, Pascual A, Pena C, Pintado V, Retamar P, Tomas M, Borges-Sa M, Garnacho-Montero J, Bou G; Study Group of Nosocomial Infections (GEIH) of the Spanish Society of Infectious Diseases, Infectious Diseases (SEIMC). Diagnosis and antimicrobial treatment of invasive infections due to multidrug-resistant Enterobacteriaceae. Guidelines of the Spanish Society of Infectious Diseases and Clinical Microbiology. Enferm Infecc Microbiol Clin. 2015 May;33(5):337.e1-337.e21. doi: 10.1016/j.eimc.2014.11.009. Epub 2015 Jan 15. PMID 25600218
- [Background] Falagas ME, Tansarli GS, Karageorgopoulos DE, Vardakas KZ. Deaths attributable to carbapenem-resistant Enterobacteriaceae infections. Emerg Infect Dis. 2014 Jul;20(7):1170-5. doi: 10.3201/eid2007.121004. PMID 24959688
- [Background] Infectious Diseases Society of America. White paper: recommendations on the conduct of superiority and organism-specific clinical trials of antibacterial agents for the treatment of infections caused by drug-resistant bacterial pathogens. Clin Infect Dis. 2012 Oct;55(8):1031-46. doi: 10.1093/cid/cis688. Epub 2012 Aug 13. PMID 22891041
- [Background] Tumbarello M, Trecarichi EM, De Rosa FG, Giannella M, Giacobbe DR, Bassetti M, Losito AR, Bartoletti M, Del Bono V, Corcione S, Maiuro G, Tedeschi S, Celani L, Cardellino CS, Spanu T, Marchese A, Ambretti S, Cauda R, Viscoli C, Viale P; ISGRI-SITA (Italian Study Group on Resistant Infections of the Societa Italiana Terapia Antinfettiva). Infections caused by KPC-producing Klebsiella pneumoniae: differences in therapy and mortality in a multicentre study. J Antimicrob Chemother. 2015 Jul;70(7):2133-43. doi: 10.1093/jac/dkv086. Epub 2015 Apr 21. PMID 25900159
- [Background] Palacios-Baena ZR, Oteo J, Conejo C, Larrosa MN, Bou G, Fernandez-Martinez M, Gonzalez-Lopez JJ, Pintado V, Martinez-Martinez L, Merino M, Pomar V, Mora-Rillo M, Rivera MA, Oliver A, Ruiz-Carrascoso G, Ruiz-Garbajosa P, Zamorano L, Bautista V, Ortega A, Morales I, Pascual A, Campos J, Rodriguez-Bano J; GEIH-GEMARA (SEIMC) and REIPI Group for CPE. Comprehensive clinical and epidemiological assessment of colonisation and infection due to carbapenemase-producing Enterobacteriaceae in Spain. J Infect. 2016 Feb;72(2):152-60. doi: 10.1016/j.jinf.2015.10.008. Epub 2015 Nov 4. PMID 26546855
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Garner JS, Jarvis WR, Emori TG, Horan TC, Hughes JM. CDC definitions for nosocomial infections, 1988. Am J Infect Control. 1988 Jun;16(3):128-40. doi: 10.1016/0196-6553(88)90053-3. PMID 2841893
- [Background] Friedman ND, Kaye KS, Stout JE, McGarry SA, Trivette SL, Briggs JP, Lamm W, Clark C, MacFarquhar J, Walton AL, Reller LB, Sexton DJ. Health care--associated bloodstream infections in adults: a reason to change the accepted definition of community-acquired infections. Ann Intern Med. 2002 Nov 19;137(10):791-7. doi: 10.7326/0003-4819-137-10-200211190-00007. PMID 12435215
- [Background] American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference: definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. Crit Care Med. 1992 Jun;20(6):864-74. PMID 1597042
- [Background] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651
- [Background] Rhee JY, Kwon KT, Ki HK, Shin SY, Jung DS, Chung DR, Ha BC, Peck KR, Song JH. Scoring systems for prediction of mortality in patients with intensive care unit-acquired sepsis: a comparison of the Pitt bacteremia score and the Acute Physiology and Chronic Health Evaluation II scoring systems. Shock. 2009 Feb;31(2):146-50. doi: 10.1097/SHK.0b013e318182f98f. PMID 18636041
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Slater A, Shann F, Pearson G; Paediatric Index of Mortality (PIM) Study Group. PIM2: a revised version of the Paediatric Index of Mortality. Intensive Care Med. 2003 Feb;29(2):278-85. doi: 10.1007/s00134-002-1601-2. Epub 2003 Jan 23. PMID 12541154
- [Background] Pang D. A relative power table for nested matched case-control studies. Occup Environ Med. 1999 Jan;56(1):67-9. doi: 10.1136/oem.56.1.67. PMID 10341749
- [Background] Stoer NC, Samuelsen SO. Inverse probability weighting in nested case-control studies with additional matching--a simulation study. Stat Med. 2013 Dec 30;32(30):5328-39. doi: 10.1002/sim.6019. Epub 2013 Oct 17. PMID 24132909
- [Background] Wolkewitz M, Beyersmann J, Gastmeier P, Schumacher M. Efficient risk set sampling when a time-dependent exposure is present: matching for time to exposure versus exposure density sampling. Methods Inf Med. 2009;48(5):438-43. doi: 10.3414/ME9241. Epub 2009 Aug 5. PMID 19657545
- [Background] Beyersmann J, Wolkewitz M, Allignol A, Grambauer N, Schumacher M. Application of multistate models in hospital epidemiology: advances and challenges. Biom J. 2011 Mar;53(2):332-50. doi: 10.1002/bimj.201000146. Epub 2011 Jan 14. PMID 21374697
- [Derived] Gutierrez-Gutierrez B, Sojo-Dorado J, Bravo-Ferrer J, Cuperus N, de Kraker M, Kostyanev T, Raka L, Daikos G, Feifel J, Folgori L, Pascual A, Goossens H, O'Brien S, Bonten MJ, Rodriguez-Bano J; EURECA project team. EUropean prospective cohort study on Enterobacteriaceae showing REsistance to CArbapenems (EURECA): a protocol of a European multicentre observational study. BMJ Open. 2017 Apr 3;7(4):e015365. doi: 10.1136/bmjopen-2016-015365. PMID 28373258
- See also: Antimicrobial resistance, global report on surveillance of World health organization — http://apps.who.int/iris/bitstream/10665/112642/1/9789241564748_eng.pdf
- See also: Surveillance report, antimicrobial resistance surveillance in Europe, ECDC. — http://ecdc.europa.eu/en/publications/Publications/antimicrobial-resistance-surveillance-europe-2013.pdf